CLINICAL TRIAL: NCT02207439
Title: A Phase II Trial of a Protease Inhibitor, Nelfinavir (NFV), Given With Definitive, Concurrent Chemoradiotherapy (CTRT) in Patients With Locally-Advanced, Human Papilloma Virus (HPV) Negative, Squamous Cell Carcinoma of the Head and Neck
Brief Title: Phase II Trial of Nelfinavir With Concurrent Chemoradiotherapy in Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 15313
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Nelfinavir; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Phase 2 (Experimental): Single Arm, Phase II study of Nelfinavir Lead-In (Period 1) Followed by Concurrent Chemoradiation with Nelfinavir (Period 2)
  Interventions: Drug: Nelfinavir (Viracept®) 1250 mg; Other: Chemoradiation

INTERVENTIONS:
Drug: Nelfinavir (Viracept®) 1250 mg — Period 1: Nelfinavir Lead-In (1250 mg bid, 7-14 days).
  Other Names: Nelfinavir Lead-In
Other: Chemoradiation — Period 2: Concurrent Chemoradiation (70 Gy over 7 weeks) with Nelfinavir (1250 mg bid)

SUMMARY:
This is a Phase II trial of definitive chemoradiotherapy (CTRT) given with the protease inhibitor,Nelfinavir (NFV), in patients with locally advanced head and neck. Eligible patients will receive a "lead-in" period of Nelfinavir (1250 mg po bid) for 7-14 days prior to initiation of CTRT. Nelfinavir will then be given concurrently with platinum-based chemotherapy and radiation therapy (planned total dose of 70 Gy over 7 weeks).

DETAILED DESCRIPTION:
This is a single-arm Phase II study of organ-preservation chemoradiotherapy given in combination with the protease inhibitor, Nelfinavir, in patients with stage II, IVa, or IVb (per AJCC version 7) squamous cell carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx. Patients start treatment with Nelfinvir at a dose of 1250 mg twice daily for 7-14 days, before continuing Nelfinvir at this dose concurrent with chemotherapy and radiation therapy (for a total dose of 70 Gy over a period of 7 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old.
* Histologically confirmed diagnosis of squamous cell carcinoma of the oral cavity, oropharynx, larynx, or hypopharynx stages III, IVa, or IVb, p16-negative on immunohistochemistry
* Determined by the treating physician to be a candidate for organ preserving, concurrent standard chemotherapy and radiation therapy to the head and neck with definitive intent.
* ECOG Performance Status 0-2
* Patients must sign an informed consent document that indicates they are aware of the investigational nature of the treatment in this protocol as well as the potential risks and benefits.
* The effects of EF5 on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, during study, until 1 month after completion of the final FMISO PET/CT scan. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Serum pregnancy testing will be required for women of childbearing potential.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria

* Prior radiation therapy to the head and neck
* Prior chemotherapy within the past 5 years
* Previous therapy with a human immunodeficiency virus (HIV) protease inhibitor
* Pregnant or lactating patients.
* Patients with known HIV disease. These patients have a high probability of treatment with anti-retroviral therapy which may interact with the nelfinavir.
* Absolute Neutrophil Count ≤ 1500 per mm3
* Platelet count ≤ 100,000 per mm3
* Serum creatinine > 1.5 times the upper limit of normal
* Serum AST or ALT > 2 times the upper limit of normal
* Serum bilirubin > 1.2 mg/dl
* Weight loss of > 10% over the past 6 months which is due to tumor wasting syndrome
* Distant metastases
* Patients receiving the following drugs that are contraindicated with NFV will be excluded: Antiarrhythmics:amiodarone, quinidine, Antimycobacterial: rifampin, Ergot Derivatives:dihydroergotamine, ergonovine, ergotamine, methylergonovine, Herbal Products: St.John's wort (hypericum perforatum), HMG-CoA Reductase Inhibitors: lovastatin,simvastatin, Neuroleptic:pimozide, Proton Pump Inhibitors, Sedative/Hypnotics: midazolam, triazolam,
* Patients receiving the following drugs will be clinically evaluated as to whether dosage/medication can be changed to permit patient on study: Anti-Convulsants: carbamazepine, Phenobarbital, Anti-Convulsant:phenytoin, Anti-Mycobacterial:rifabutin, PDE5 Inhibitors: sildenafil, vardenafil, tadalafil, HMG-CoA: Reductase Inhibitors: atorvastatin, rosuvastatin, Immuno-suppressants: cyclosporine,tacrolimus, sirolimus, Narcotic Analgesic: methadone, Oral Contraceptive:ethinyl estradiol, Macrolide Antibiotic:azithromycin, Inhaled/nasal steroid fluticasone, Antidepressant: trazodone.
* Women of childbearing potential who have a positive result on screening urine pregnancy test.
* Subjects with moderate-severe renal disease.
* History of allergic reactionsattributed to Flagyl (metronidazole), which has a chemical structure similar to FMISO.
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2022-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lin, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm, 2 Period, Phase 2 Trial: Period 1: Nelfinavir Lead-In (1250 mg bid, 7-14 days)
  Period 2: Definitive Chemoradiotherapy with Nelfinavir (70 Gy radiotherapy over 7 weeks)
Period: Nelfinavir Lead-In
Arm/Group | Single Arm, 2 Period, Phase 2 Trial
Started | 17
Completed | 17
Not Completed | 0
Period: Chemoradiotherapy With Nelfinavir
Arm/Group | Single Arm, 2 Period, Phase 2 Trial
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Phase 2: Nelfinavir (Viracept®) 1250 mg
  FMISO
Arm/Group | Single Arm Phase 2
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 61 [43 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17
Locoregional head and neck cancer [Number; unit: participants] | 17

OUTCOME MEASURES:

1. Primary Outcome: Locoregional Control
Description: locoregional control determined via diagnostic imaging and clinical examination.
Time Frame: 5 years
Measure: Number (64.7% Confidence Interval); unit: participants
Groups:
- Single Arm Phase 2: Locoregional Control
Arm/Group | Single Arm Phase 2
Number analyzed (Participants) | 17
participants | 17 [11 to 17]

2. Secondary Outcome: Decrease in Hypoxia From Nelfinavir
Description: Decrease in Hypoxia from Nelfinavir was determined by change in uptake and volume as assessed via 18f-FMISO or 18f-EF5 PET/CT pre-Nelfinavir versus post Nelfnavir lead-in
Time Frame: 7-14 days
Measure: Number (67% Confidence Interval); unit: participants
Arm/Group | Single Arm, 2 Period, Phase 2 Trial
Number analyzed (Participants) | 12
participants | 12 [8 to 12]

3. Secondary Outcome: Change in Glucose Metabolism From Nelfinavir
Description: Change in Glucose Metabolism from Nelfinavir was determined by change in glucose uptake as assessed via FDG-PET/CT pre-Nelfinavir versus post Nelfnavir lead-in
Time Frame: From the initiation of any study procedures to 30 days following the completion of 7 chemoradiation
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm, 2 Period, Phase 2 Trial
Number analyzed (Participants) | 17
Participants | 17

ADVERSE EVENTS:
Time Frame: Start: at initiation of first study procedure (baseline PET/CT imaging) Ends: 30 days after last day of chemoradiation
Arm/Group | Single Arm Phase 2
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 17/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Phase 2 (N=17)
Dysgeusia (Nervous system disorders) | 1 (1) — A disorder characterized by abnormal sensual experience with the taste of foodstuffs; it can be related to a decrease in the sense of smell.
Allergic reaction (Immune system disorders) | 1 (1) — A disorder characterized by an adverse local or general response from exposure to an allergen.
Anemia (Blood and lymphatic system disorders) | 1 (1) — A disorder characterized by an reduction in the amount of hemoglobin in 100 ml of blood.
Anorexia (Metabolism and nutrition disorders) | 2 (2) — A disorder characterized by a loss of appetite.
Aspartate aminotransferase increased (Investigations) | 1 (1) — A finding based on laboratory test results that indicate an increase in the level of aspartate aminotransferase (AST or SGOT) in a blood specimen.
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (5) — A disorder characterized by inhalation of solids or liquids into the lungs.
Cholecystitis (Hepatobiliary disorders) | 1 (1) — A disorder characterized by inflammation involving the gallbladder. It may be associated with the presence of gallstones.
Dysphagia (Gastrointestinal disorders) | 2 (2) — A disorder characterized by difficulty in swallowing.
Esophagitis (Gastrointestinal disorders) | 1 (1) — A disorder characterized by inflammation of the esophageal wall.
Headache (Nervous system disorders) | 1 (1) — A disorder characterized by a sensation of marked discomfort in various parts of the head, not confined to the area of distribution of any nerve.
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — A disorder characterized by laboratory test results that indicate an elevation in the concentration of blood sugar.
Hypertension (Vascular disorders) | 1 (1) — A disorder characterized by a pathological increase in blood pressure
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) — A disorder characterized by laboratory test results that indicate a low concentration of potassium in the blood.
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) — A disorder characterized by laboratory test results that indicate a low concentration of sodium in the blood.
Lymphocyte count decreased (Investigations) | 5 (9) — A finding based on laboratory test results that indicate a decrease in number of lymphocytes in a blood specimen.
Mucositis oral (Gastrointestinal disorders) | 3 (3) — A disorder characterized by inflammation of the oral mucosal.
Neutrophil count decreased (Investigations) | 1 (3) — A finding based on laboratory test results that indicate a decrease in number of neutrophils in a blood specimen.
Platelet count decreased (Investigations) | 1 (2) — A finding based on laboratory test results that indicate a decrease in number of platelets in a blood specimen.
Sinus bradycardia (Cardiac disorders) | 1 (1) — A disorder characterized by a dysrhythmia with a heart rate less than 60 beats per minute that originates in the sinus node.
White blood cell decreased (Investigations) | 1 (46) — A finding based on laboratory test results that indicate an decrease in number of white blood cells in a blood specimen.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Phase 2 (N=17)
Agitation (Psychiatric disorders) | 1 (1) — A disorder characterized by a state of restlessness associated with unpleasant feelings of irritability and tension.
Alanine aminotransferase increased (Investigations) | 3 (4) — A finding based on laboratory test results that indicate an increase in the level of alanine aminotransferase (ALT or SGPT) in the blood specimen.
Alkaline phosphatase increased (Investigations) | 2 (2) — A finding based on laboratory test results that indicate an increase in the level of alkaline phosphatase in a blood specimen.
Allergic reaction (Immune system disorders) | 1 (1) — A disorder characterized by an adverse local or general response from exposure to an allergen.
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) — A disorder characterized by a decrease in density of hair compared to normal for a given individual at a given age and body location
Anemia (Blood and lymphatic system disorders) | 8 (17) — A disorder characterized by an reduction in the amount of hemoglobin in 100 ml of blood.
Anorexia (Metabolism and nutrition disorders) | 9 (17) — A disorder characterized by a loss of appetite.
Anxiety (Psychiatric disorders) | 3 (4) — A disorder characterized by apprehension of danger and dread accompanied by restlessness, tension, tachycardia, and dyspnea unattached to a clearly identifiable stimulus.
Aspartate aminotransferase increased (Investigations) | 1 (1) — A finding based on laboratory test results that indicate an increase in the level of aspartate aminotransferase (AST or SGOT) in a blood specimen.
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) — A disorder characterized by inhalation of solids or liquids into the lungs.
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — A disorder characterized by marked discomfort sensation in the back region.
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — A disorder characterized by inflammation of the skin characterized by the presence of bullae which are filled with fluid.
Constipation (Gastrointestinal disorders) | 8 (9) — A disorder characterized by irregular and infrequent or difficult evacuation of the bowels.
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) — A disorder characterized by sudden, often repetitive, spasmodic contraction of the thoracic cavity, resulting in violent release of air from the lungs and usually accompanied by a distinctive sound.
Creatinine increased (Investigations) | 2 (2) — A finding based on laboratory test results that indicate increased levels of creatinine in a biological specimen.
Dehydration (Metabolism and nutrition disorders) | 2 (2) — A disorder characterized by excessive loss of water from the body. It is usually caused by severe diarrhea, vomiting or diaphoresis.
Depression (Psychiatric disorders) | 2 (2) — A disorder characterized by melancholic feelings of grief or unhappiness.
Dermatitis radiation (Injury, poisoning and procedural complications) | 14 (21) — A finding of cutaneous inflammatory reaction occurring as a result of exposure to biologically effective levels of ionizing radiation.
Diarrhea (Gastrointestinal disorders) | 8 (8) — A disorder characterized by frequent and watery bowel movements.
Dizziness (Nervous system disorders) | 3 (3) — A disorder characterized by a disturbing sensation of lightheadedness, unsteadiness, giddiness, spinning or rocking.
Dry mouth (Gastrointestinal disorders) | 8 (8) — A disorder characterized by reduced salivary flow in the oral cavity.
Dysgeusia (Nervous system disorders) | 15 (22) — A disorder characterized by abnormal sensual experience with the taste of foodstuffs; it can be related to a decrease in the sense of smell.
Dysphagia (Gastrointestinal disorders) | 11 (17) — A disorder characterized by difficulty in swallowing.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — A disorder characterized by an uncomfortable sensation of difficulty breathing.
Ear pain (Ear and labyrinth disorders) | 1 (1) — A disorder characterized by a sensation of marked discomfort in the ear.
Edema face (General disorders) | 1 (1) — A disorder characterized by swelling due to excessive fluid accumulation in facial tissues.
Edema limbs (General disorders) | 2 (2) — A disorder characterized by swelling due to excessive fluid accumulation in the upper or lower extremities.
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4 (4) — A disorder characterized by target lesions (a pink-red ring around a pale center).
Esophageal pain (Skin and subcutaneous tissue disorders) | 1 (2) — A disorder characterized by a sensation of marked discomfort in the esophageal region.
Fatigue (General disorders) | 11 (17) — A disorder characterized by a state of generalized weakness with a pronounced inability to summon sufficient energy to accomplish daily activities.
Fever (General disorders) | 2 (3) — A disorder characterized by elevation of the body's temperature above the upper limit of normal.
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) — A disorder characterized by reflux of the gastric and/or duodenal contents into the distal esophagus.
Gastroparesis (Gastrointestinal disorders) | 1 (1) — A disorder characterized by an incomplete paralysis of the muscles of the stomach wall resulting in delayed emptying of the gastric contents into the small intestine.
Headache (Nervous system disorders) | 2 (2) — A disorder characterized by a sensation of marked discomfort in various parts of the head, not confined to the area of distribution of any nerve.
Hemorrhoids (Gastrointestinal disorders) | 1 (1) — A disorder characterized by the presence of dilated veins in the rectum and surrounding area.
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) — A disorder characterized by repeated gulp sounds that result from an involuntary opening and closing of the glottis. This is attributed to a spasm of the diaphragm.
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) — A disorder characterized by harsh and raspy voice arising from or spreading to the larynx.
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) — A disorder characterized by laboratory test results that indicate an elevation in the concentration of blood sugar.
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) — A disorder characterized by laboratory test results that indicate an elevation in the concentration of potassium in the blood; associated with kidney failure or sometimes with the use of diuretic drugs.
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) — A disorder characterized by laboratory test results that indicate a low concentration of albumin in the blood.
Hypocalcemia (Metabolism and nutrition disorders) | 4 (6) — A disorder characterized by laboratory test results that indicate a low concentration of calcium in the blood.
Hypokalemia (Metabolism and nutrition disorders) | 2 (5) — A disorder characterized by laboratory test results that indicate a low concentration of potassium in the blood.
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (6) — A disorder characterized by laboratory test results that indicate a low concentration of magnesium in the blood.
Hyponatremia (Metabolism and nutrition disorders) | 5 (8) — A disorder characterized by laboratory test results that indicate a low concentration of sodium in the blood.
Hypotension (Vascular disorders) | 1 (1) — A disorder characterized by a blood pressure that is below the normal expected for an individual in a given environment.
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — A disorder characterized by swelling due to an excessive accumulation of fluid in the larynx.
Localized edema (General disorders) | 1 (2) — A disorder characterized by swelling due to excessive fluid accumulation at a specific anatomic site.
Lymphocyte count decreased (Investigations) | 2 (2) — A finding based on laboratory test results that indicate a decrease in number of lymphocytes in a blood specimen.
Lymphocyte count increased (Investigations) | 1 (1) — A finding based on laboratory test results that indicate an abnormal increase in the number of lymphocytes in the blood, effusions or bone marrow.
Middle ear inflammation (Ear and labyrinth disorders) | 1 (2) — A disorder characterized by inflammation (physiologic response to irritation), swelling and redness to the middle ear.
Mucositis oral (Gastrointestinal disorders) | 9 (13) — A disorder characterized by inflammation of the oral mucosal.
Nausea (Gastrointestinal disorders) | 7 (7) — A disorder characterized by a queasy sensation and/or the urge to vomit.
Neck edema (General disorders) | 7 (8) — A disorder characterized by swelling due to an accumulation of excessive fluid in the neck.
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) — A disorder characterized by marked discomfort sensation in the neck area.
Oral pain (Gastrointestinal disorders) | 3 (3) — A disorder characterized by a sensation of marked discomfort in the mouth, tongue or lips.
Pain (General disorders) | 5 (8) — A disorder characterized by the sensation of marked discomfort, distress or agony.
Platelet count decreased (Investigations) | 2 (5) — A finding based on laboratory test results that indicate a decrease in number of platelets in a blood specimen.
Prostatic pain (Reproductive system and breast disorders) | 1 (1) — A disorder characterized by a sensation of marked discomfort in the prostate gland.
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) — A disorder characterized by the presence of macules (flat) and papules (elevated)
Salivary duct inflammation (Gastrointestinal disorders) | 10 (14) — A disorder characterized by inflammation of the salivary duct.
Somnolence (Nervous system disorders) | 1 (1) — A disorder characterized by characterized by excessive sleepiness and drowsiness.
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) — A disorder characterized by of marked discomfort in the throat
Stomach pain (Gastrointestinal disorders) | 1 (1) — A disorder characterized by a sensation of marked discomfort in the stomach.
Thromboembolic event (Vascular disorders) | 1 (1) — A disorder characterized by occlusion of a vessel by a thrombus that has migrated from a distal site via the blood stream.
Tinnitus (Ear and labyrinth disorders) | 3 (3) — A disorder characterized by noise in the ears, such as ringing, buzzing, roaring or clicking.
Tremor (Nervous system disorders) | 3 (3) — A disorder characterized by the uncontrolled shaking movement of the whole body or individual parts.
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 6 (7) — A disorder characterized by a change in the sound and/or speed of the voice.
Vomiting (Gastrointestinal disorders) | 2 (2) — A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth.
Weight loss (Investigations) | 4 (6) — A finding characterized by a decrease in overall body weight; for pediatrics, less than the baseline growth curve.
White blood cell decreased (Investigations) | 17 (332) — A finding based on laboratory test results that indicate an decrease in number of white blood cells in a blood specimen.
Infections and infestations (Infections and infestations) | 2 (3) — Infections and infestations
Investigations (Investigations) | 2 (8) — Investigations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT02207439/Prot_SAP_000.pdf